CLINICAL TRIAL: NCT05800054
Title: Effect of NST Whole-course Nutritional Management on Nutritional Status and Adverse Reactions in Patients With Esophageal Cancer Undergoing Concurrent Chemoradiotherapy
Brief Title: Effect of NST Whole-course Nutritional Management on Nutritional Status and Adverse Reactions in Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GXL-001
Record Dates: First submitted 2022-08-14; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Neoplasms; Adverse Drug Event
MeSH Terms: conditions — Esophageal Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Docetaxel; Drug Therapy; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NST intervenes throughout the process (Experimental): 1. Nutritionists formulate nutritional programs and manage them in a refined manner.
     The nutritionist urges the patient to report daily to ensure that the patient's energy and protein are in place
  2. Radiotherapy
  3. chemotherapy
  Interventions: Dietary Supplement: Nutritional Support Team; Drug: Docetaxel; Drug: cisplatin; Radiation: Radiotherapy
- Routine nutrition guidance group for esophageal cancer (Experimental): 1. Patients perform their own nutrition regimen, and the nutritionist is not involved in management
  2. Radiotherapy
  3. chemotherapy
  Interventions: Drug: Docetaxel; Drug: cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Dietary Supplement: Nutritional Support Team — Nutritionists formulate nutritional programs and manage them in a refined manner. On the basis of the patient's natural diet (food and homogenate meal), enteral nutritional preparations or parenteral nutritional supplements are given according to the patient's gastrointestinal obstruction, dietary structure, and food intake. Energy 30-35kcal/kg/d, protein 1.2-1.5g/kg/d. Enteral nutrition administration route: oral or tube feeding or ostomy, oral feeding is preferred; severe obstruction of eating or oral intake cannot meet the target nutrition, choose tube feeding or ostomy. When it is expected that enteral nutrition cannot meet 60% of the target energy requirement for 3 to 5 days, choose parenteral nutrition. The enteral nutritional preparation adopts the whole protein enteral nutritional preparation Nengquan, and/or the tumor nutritional preparation Ruineng, and/or whey protein powder.
  Other Names: taixinsheng
  Arms: NST intervenes throughout the process
Drug: Docetaxel — 60-75 mg/m2, d1, at least 2 cycles in parallel with radiotherapy
  Other Names: chemotherapy
Drug: cisplatin — cisplatin 25mg/m2 d1-3, 21-28d/cycle. at least 2 cycles in parallel with radiotherapy
  Other Names: chemotherapy
Radiation: Radiotherapy — image-guided intensity-modulated radiotherapy (IGRT) or intensity-modulated radiotherapy (IMRT); Irradiation targets include primary lesions, clinical targets, positive lymph nodes, and lymph node drainage areas. Dose splitting/prescription dose, 95% volume PGTV-T60-66Gy/30-35 times, PGTV-N 60-66Gy/30-35 times, PCTV-T 46-50Gy/23-25 times, PCTV-N46-50Gy/23-25 times.

SUMMARY:
This study is a randomized, open, parallel controlled clinical trial. The main purpose of this study was to compare the changes in body weight/body mass index (BMI) before and after treatment between the two groups of patients with NST full-course nutritional management and without NST full-course nutritional management.

The secondary objective was to compare the quality of life, nutritional status, immune function and inflammatory response, adverse reactions of radiotherapy and chemotherapy, and short-term/long-term efficacy between the two groups.

The treatment plan was: esophageal cancer with routine nutrition guidance as the control group, and the NST whole-process intervention guidance as the experimental group.

1. Experimental group: NST whole-course intervention

1. Nutritionists formulate nutritional programs and manage them in a refined manner. On the basis of the patient's natural diet (food and homogenate meal), enteral nutritional preparations or parenteral nutritional supplements are given according to the patient's gastrointestinal obstruction, dietary structure, and food intake. Energy 30-35kcal/kg/d, protein 1.2-1.5g/kg/d. Enteral nutrition administration route: oral or tube feeding or ostomy, oral feeding is preferred; severe obstruction of eating or oral can not meet the target nutrition, choose tube feeding or ostomy. When it is expected that enteral nutrition cannot meet 60% of the target energy requirement for 3 to 5 days, choose parenteral nutrition. The enteral nutritional preparation adopts the whole protein enteral nutritional preparation Nengquan, and/or the tumor nutritional preparation Ruineng, and/or whey protein powder.
2. Radiotherapy
3. Chemotherapy 2. Control group: routine nutrition guidance for esophageal cancer

(1) Nutritional therapy: The nutritional program was the same as that of the experimental group, and the patients performed it themselves.

(2) Concurrent chemoradiotherapy: the same as the experimental group.

Efficacy evaluation:

1. Body weight and body mass index (BMI)
2. Quality of life score (EORTCQLQ-C30)
3. Nutritional status
4. Immune function and inflammatory response (total lymphocytes, CRP, IL-6)

(4) Intestinal mucosal barrier and intestinal flora (5) Adverse reactions of radiotherapy and chemotherapy (6) Short-term/long-term efficacy (5) Evaluation of treatment side effects (6) Short-term/long-term efficacy

DETAILED DESCRIPTION:
This study is a randomized, open, parallel controlled clinical trial. The main purpose of this study was to compare the changes in body weight/body mass index (BMI) before and after treatment between the two groups of patients with NST full-course nutritional management and without NST full-course nutritional management.

The secondary objective was to compare the quality of life, nutritional status, immune function and inflammatory response, adverse reactions of radiotherapy and chemotherapy, and short-term/long-term efficacy between the two groups.

The treatment plan was: esophageal cancer with routine nutrition guidance as the control group, and the NST whole-process intervention guidance as the experimental group.

1. Experimental group: NST whole-course intervention

1. Nutritionists formulate nutritional programs and manage them in a refined manner. On the basis of the patient's natural diet (food and homogenate meal), enteral nutritional preparations or parenteral nutritional supplements are given according to the patient's gastrointestinal obstruction, dietary structure, and food intake. Energy 30-35kcal/kg/d, protein 1.2-1.5g/kg/d. Enteral nutrition administration route: oral or tube feeding or ostomy, oral feeding is preferred; severe obstruction of eating or oral can not meet the target nutrition, choose tube feeding or ostomy. When it is expected that enteral nutrition cannot meet 60% of the target energy requirement for 3 to 5 days, choose parenteral nutrition. The enteral nutritional preparation adopts the whole protein enteral nutritional preparation Nengquan, and/or the tumor nutritional preparation Ruineng, and/or whey protein powder.

   Enteral nutrition preparations should choose Nengquan, and the dose of Nengjian: (a) No/mild obstruction, can eat ordinary diet, the food intake is not reduced or less than 1/3 before the disease, and 10-15kcal of Nengjian is given. /kg/d; (b) moderate obstruction, can eat soft food, the food intake is less than 1/3~2/3 before the disease, and can give 15-20kcal/kg/d; (c) severe obstruction, can not Eating, the food intake is reduced by >= 2/3 compared with that before the disease, and can be given 20-25kcal/kg/d of all-vegetarian food; Dosage of whey protein powder: (a) albumin 35~40g/L, supplemented with whey protein powder 10g; (b) albumin 30~35g/L, supplemented with whey protein powder 20g; (c) albumin <30g /L, supplement whey protein powder 30g.

   Nutritionists urge patients to report daily to ensure adequate energy and protein supplementation.
2. Radiotherapy: image-guided intensity-modulated radiotherapy (IGRT) or intensity-modulated radiotherapy (IMRT); the irradiation target areas include primary lesions, clinical target areas, positive lymph nodes, and lymph node drainage areas. Dose split/prescribed dose, 95% volume PGTV-T60-66Gy/30-35 times, PGTV-N 60-66Gy/30-35 times, PCTV-T 46-50Gy/23-25 times, PCTV-N46-50Gy/ 23-25 times.
3. Chemotherapy: Docetaxel 60-75mg/m2, d1, DDP 25mg/m2 d1-3, 21-28d/cycle. Simultaneous with radiotherapy for at least 2 cycles, after radiotherapy, the choice of whether to continue adjuvant chemotherapy is based on specific circumstances.

2. Control group: routine nutrition guidance for esophageal cancer

1. Nutritional therapy: The nutritional program was the same as that of the experimental group, and the patients performed it themselves.
2. Concurrent chemoradiotherapy: the same as the experimental group.

Efficacy evaluation:

1. Body weight and body mass index (BMI)
2. Quality of life score (EORTCQLQ-C30)
3. Nutritional status
4. Immune function and inflammatory response (total lymphocytes, CRP, IL-6)

(4) Intestinal mucosal barrier and intestinal flora (5) Adverse reactions of radiotherapy and chemotherapy (6) Short-term/long-term efficacy (5) Evaluation of treatment side effects (6) Short-term/long-term efficacy Statistical methods: All statistical tests were two-sided, and P values < 0.05 were considered statistically significant. Data are presented as x ±s. Quantitative data were analyzed by t test and variance analysis, qualitative data were analyzed by X2 test, and survival data were analyzed by Kaplan Meire method, logrank test, and Cox regression.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent; must have good compliance with the treatment plan and follow-up.
* No gender restriction, but age between 18 and 75 years old;
* Cytological or histological is confirmed esophageal squamous cell carcinoma;
* Non-surgical treatment of stage II-III primary esophageal cancer (except biopsy);
* The primary tumor can be evaluated;
* No distant organ metastasis;
* PG-SGA score B (2~8) or C (≥9);
* KPS score ≥ 70 points, ECOG physical condition score 0-1 points;
* The function of major organs (bone marrow, liver, kidney function) 7 days before treatment, meet the following criteria: Blood routine examination standards (without blood transfusion within 14 days):

  * Hemoglobin (HB) ≥ 100g/L;

    * White blood cells (WBC) ≥ 4×109/L; Absolute neutrophil count (ANC) ≥1.5×109/L;

      * Platelet (PLT) ≥ 100×109/L.
* The biochemical examination shall meet the following standards:

  * Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);

    * Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 1.5 times ULN;

      * Serum creatinine (Cr) ≤ 1.5 times ULN or creatinine clearance rate (CCr) ≥ 60ml/min.
* Expected survival ≥ 6 months.

Exclusion Criteria:

* No malnutrition or nutritional risk; PG-SGA score of A;
* Severely impaired intestinal function, or intolerance of enteral nutrition;
* Severe vomiting, gastrointestinal bleeding, intestinal obstruction;
* Patients with very severe malnutrition cannot tolerate radiotherapy and chemotherapy;
* The primary tumor or lymph node has received radiotherapy, chemotherapy or targeted therapy;
* Suffering from other malignant tumors within 5 years (except for completely cured cervical carcinoma in situ or skin basal cell carcinoma);
* Subjects who have received other drug trials within the past month;
* Those with severe allergic history or idiosyncratic constitution;
* Those with a history of severe lung or heart disease;
* Serious comorbidities, such as uncontrolled hypertension, heart failure, etc.;
* Pregnant or breastfeeding women;
* Currently or planning to participate in other clinical trials;
* Refusal or inability to sign the informed consent form to accept participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight and body mass index (BMI) | up to 3 years
  BMI = weight ÷ height2. (Unit of weight: kg; Height unit: meters),During treatment: Body weight was recorded daily and BMI was recorded weekly,BMI values are recorded every Friday

SECONDARY OUTCOMES:
Quality of life score | up to 3 years
  EORTCQLQ-C30，EORTC:The European O-rganization for Reasearch and Treatment of Cancer)，QOL-C30 (Quality of Life Questionnare-Core 30，Assessments are conducted every two weeks on Fridays of the second week
hemoglobin | up to 3 years
  Compare the numerical changes of hemoglobin every two weeks
serum albumin | up to 3 years
  Compare the numerical changes of serum albumin every two weeks
ORR | through study completion, an average of 36 month
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No